## UniSZA-PTPIP-42-GP 001-BR 008(01)



Jawatankuasa Etika Penyelidikan Manusia UniSZA I UniSZA Human Research Ethics Committee (UHREC)

Acute Effect of Melon Manis Terengganu Peel Powder on Glycemic Response, Satiety, and Food Intake in Adults at Risk for Type 2 Diabetes

1 March 2022



## INFORMED CONSENT FORM

| Research | Title: Ad | cute eff | ect of hi | gh fibe | er powde | r developed | from | Melon | Manis | Terengganu | peel | on |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| glycemic re | esponse, | satiety | and foo | d intak | e in adult | s at risk for | type 2 | 2 diabet | es | | | |

## **\Name of Principal Investigator/ (MMC No.)\*:**

1. Ms Ong Ying Qian

## Name of co-Researcher(s)/ (MMC No.)\*:

- 1. Prof Dr Sakinah Harith
- 2. Prof Madya Dr Mohd Razif Shahril
- 3. Dr Norshazila Shahidan
- 4. Prof Madya Dr Hermizi Hapidin

To become a participant of this research, you or your legal representative (parent/ guardian) must sign this form.

By signing this page, I am confirming the following:

- I have read the Research Information Sheet (UniSZA-PTPIP-42-GP 001-BR 006(01) and this Informed Consent Form, or it has been read to me.
- I understand the nature and scope of research being undertaken including any information regarding the risk in this research and I have had time to think about it.
- All my questions relating to this research and my participation therein have been answered to my satisfaction.
- I voluntarily agree to take part in this research, to follow the study procedures and to provide all necessary information to the investigators as requested.
- I may at any time choose to withdraw from this research without giving any reasons.
- Except for damages resulting from negligent or malicious conduct of the researcher(s), I hereby release and discharge Universiti Sultan Zainal Abidin and all the participating researchers from all liability associated with, arising out of, or related to my participation and agree to hold them harmless from any harm or loss that may be incurred by me due to my participation in the research.
- I have received a copy of the Research Information Sheet (UniSZA-PTPIP-42-GP 001-BR 006(01).

| Participant Name: | Participant I.C No/ Passport No. |
|---|---|
| Signature/ Thumb Print of Participant/ Legal Representative: | Date: |

| Name of Individual Conducting Consent Discussion: | Role: | |
|---|---|---|
| Ms Ong Ying Qian | Researcher/ Research Assistant | t/ |
| | Enumerator/ Field Assistant | t/ |
| | Others (please specify) | |

<sup>\*</sup>To be included if applicable



| Signature of Individual Conducting Consent Discussion: | Date: |
|--------------------------------------------------------|-------|

**Note:** All participants who are involved in this study will not be covered by insurance.